CLINICAL TRIAL: NCT05303220
Title: A Phase 1, Open-label, Randomized, Crossover Study to Evaluate the Bioavailability of Branebrutinib in a Tablet Formulation Relative to Branebrutinib (RBA) in a Capsule Formulation Including the Effect of Food (Low-fat/Low-calorie and a High-fat/High-calorie) on the Bioavailability of Branebrutinib From a Tablet Formulation and a Double-blind Study to Evaluate the Safety and Pharmacokinetics of Branebrutinib From a Tablet Formulation in a Multiple-dose Arm in Healthy Participants
Brief Title: A Study to Assess Relative Bioavailability of Branebrutinib, From a Tablet Formulation to the Capsule Formulation, the Effect of Food on the Bioavailability of Branebrutinib From a Tablet Formulation, and the Safety and Drug Levels of Branebrutinib From a Tablet Formulation in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM014-036; 2015-004300-38 (EudraCT Number)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — branebrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1 Treatment A (Experimental)
  Interventions: Drug: Branebrutinib
- Part 1 Treatment B (Experimental)
  Interventions: Drug: Branebrutinib
- Part 1 Treatment C (Experimental)
  Interventions: Drug: Branebrutinib
- Part 1 Treatment D (Experimental)
  Interventions: Drug: Branebrutinib
- Part 2 Treatment A (Experimental)
  Interventions: Drug: Branebrutinib
- Part 2 Treatment B (Experimental)
  Interventions: Drug: Branebrutinib
- Part 2 Treatment C (Experimental)
  Interventions: Drug: Branebrutinib
- Part 3 Treatment A (Experimental)
  Interventions: Drug: Branebrutinib
- Part 3 Treatment B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Branebrutinib — Specified dose on specified days
  Other Names: BMS-986195
  Arms: Part 1 Treatment A; Part 1 Treatment B; Part 1 Treatment C; Part 1 Treatment D; Part 2 Treatment A; Part 2 Treatment B; Part 2 Treatment C; Part 3 Treatment A
Drug: Placebo — Specified Dose on specified days
  Arms: Part 3 Treatment B

SUMMARY:
The purpose of this study is to assess the relative bioavailability of branebrutinib tablet formulation relative to the capsule formulation in order to identify doses that would provide exposures similar to the capsule formulation over the dose range that may be used in future clinical studies, evaluate the effect of food on the bioavailability of branebrutinib from a tablet formulation at a dose projected to provide similar pharmacokinetics (PK) as the 9 mg capsule formulation, and evaluate the safety and the PK of multiple oral dose of tablet formulation of branebrutinib in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants, of any race, as determined by no deviation considered significant by the investigator from normal in medical history, physical examination, 12-lead ECG measurements, and clinical laboratory determinations at screening or at check-in
* Body mass index (BMI) 18.0 to 33.0 kg/m2, inclusive. BMI = weight (kg)/(height [m])2 for participants
* Participant is afebrile (febrile is defined as ≥ 38°C or ≥100.4°F), with systolic blood pressure ≥ 90 and ≤ 160 mm Hg, diastolic blood pressure ≥ 50 and ≤ 100 mm Hg, and pulse rate ≥ 40 and ≤ 100 beats per minute at screening

Exclusion Criteria:

* Any significant acute or chronic medical illness that presents a potential risk to the participant in the opinion of the investigator and/or may compromise the objectives of the study
* History of clinically significant endocrine, gastrointestinal (GI), cardiovascular (CV), peripheral vascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary (GU) abnormalities/diseases
* History of acute or chronic bacterial, fungal, or viral infection necessitating treatment or inpatient admission within the 3 months prior to screening, or active/symptomatic infection at the time of screening

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 14
Area under the plasma concentration-time curve (AUC) from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to Day 14
AUC from time zero extrapolated to infinite time (AUC(INF)) | Up to Day 14
Number of participants with adverse events (AEs) | Up to 30 days post last scheduled visit
Number of participants with vital sign abnormalities | Up to Day 14
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 14
Number of participants with physical examination abnormalities | Up to Day 14
Number of participants with clinical laboratory abnormalities | Up to Day 14

SECONDARY OUTCOMES:
Geometric mean ratio of Cmax | Up to Day 17
Geometric mean ratio of AUC(0-T) | Up to Day 17
Geometric mean ratio of AUC(INF) | Up to Day 17
Time of maximum observed plasma concentration (Tmax) | Up to Day 17
Apparent total body clearance (CLT/F) | Up to Day 14
Apparent volume of distribution (Vz/F) | Up to Day 14
Number of participants with AEs | Up to 30 days post last scheduled visit
Number of participants with vital sign abnormalities | Up to Day 14
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 14
Number of participants with physical examination abnormalities | Up to Day 14
Number of participants with clinical laboratory abnormalities | Up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Miami, Florida, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm